CLINICAL TRIAL: NCT00623610
Title: Beta-Cell Transplantation in Pre-Uremic Patients With Type 1 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AZ-VUB (Other)
Collaborators: Vrije Universiteit Brussel (Other); Universitaire Ziekenhuizen KU Leuven (Other); Universiteit Antwerpen (Other); Erasme University Hospital (Other)
Responsible Party: Bart Keymeulen, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BK-Tx-04
Record Dates: First submitted 2008-02-19; First posted 2008-02-26 (Estimated); Last update posted 2008-02-26 (Estimated); Status verified 2008-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes mellitus, type 1; pancreatic beta cell; transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: islet cell grafts — Intraportal injection of an islet cell graft into the liver.

SUMMARY:
To examine whether temporary immunosuppression with ATG, tacrolimus and MMF allows prolonged survival of beta cell allografts in type 1 diabetic patients with early chronic complications of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* type 1 insulin-dependent diabetic patients in relatively good general condition
* non-smoker
* body weight < 80 kg
* C-peptide < 0.03 nmol/l (<0.09 µg/l) 6 min. after glucagon IV (1mg) (glycemia > 180 mg/dl)
* EBV antibody positive
* cooperative and reliable patient giving informed consent by signature; the patient should be informed in sufficient detail on the content and procedure of the protocol, indicating potential risks of intervention and of immunosuppressive therapy; the patient should also be informed that withdrawal of immunosuppressive therapy in patients with persistent plasma C-peptide positivity may result in subsequent loss of ß-cell graft function; the ß cell implant should be identified as a clinical trial

Exclusion Criteria:

* history of thrombosis or pulmonary embolism
* abnormal liver function
* HLA antibodies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2000-09; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Evidence of clinically relevant beta cell function. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bart Keymeulen, MD, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (2):
- Belgium (2):
  - Universitair Ziekenhuis and Diabetes Research Center - Brussels Free University-VUB, Brussels
  - Department of Endocrinology and Nephrology, UZ Gasthuisberg, Katholieke Universiteit Leuven -KUL, Leuven

REFERENCES:
- [Background] Movahedi B, Keymeulen B, Lauwers MH, Goes E, Cools N, Delvaux G. Laparoscopic approach for human islet transplantation into a defined liver segment in type-1 diabetic patients. Transpl Int. 2003 Mar;16(3):186-90. doi: 10.1007/s00147-002-0517-7. Epub 2003 Feb 15. PMID 12664214
- [Background] Maleux G, Gillard P, Keymeulen B, Pipeleers D, Ling Z, Heye S, Thijs M, Mathieu C, Marchal G. Feasibility, safety, and efficacy of percutaneous transhepatic injection of beta-cell grafts. J Vasc Interv Radiol. 2005 Dec;16(12):1693-7. doi: 10.1097/01.RVI.0000182506.88739.39. PMID 16371537
- [Result] Keymeulen B, Gillard P, Mathieu C, Movahedi B, Maleux G, Delvaux G, Ysebaert D, Roep B, Vandemeulebroucke E, Marichal M, In 't Veld P, Bogdani M, Hendrieckx C, Gorus F, Ling Z, van Rood J, Pipeleers D. Correlation between beta cell mass and glycemic control in type 1 diabetic recipients of islet cell graft. Proc Natl Acad Sci U S A. 2006 Nov 14;103(46):17444-9. doi: 10.1073/pnas.0608141103. Epub 2006 Nov 7. PMID 17090674
- [Derived] Lee D, Gillard P, Hilbrands R, Ling Z, Van de Velde U, Jacobs-Tulleneers-Thevissen D, Maleux G, Lapauw B, Crenier L, De Block C, Mathieu C, Pipeleers D, Keymeulen B. Use of Culture to Reach Metabolically Adequate Beta-cell Dose by Combining Donor Islet Cell Isolates for Transplantation in Type 1 Diabetes Patients. Transplantation. 2020 Oct;104(10):e295-e302. doi: 10.1097/TP.0000000000003321. PMID 32433237
- [Derived] Balke EM, Demeester S, Lee D, Gillard P, Hilbrands R, Van de Velde U, Van der Auwera BJ, Ling Z, Roep BO, Pipeleers DG, Keymeulen B, Gorus FK. SLC30A8 polymorphism and BMI complement HLA-A*24 as risk factors for poor graft function in islet allograft recipients. Diabetologia. 2018 Jul;61(7):1623-1632. doi: 10.1007/s00125-018-4609-z. Epub 2018 Apr 20. PMID 29679103
- [Derived] Lee D, Keymeulen B, Hilbrands R, Ling Z, Van de Velde U, Jacobs-Tulleneers-Thevissen D, Maleux G, Lapauw B, Crenier L, De Block C, Mathieu C, Pipeleers D, Gillard P. Age and Early Graft Function Relate With Risk-Benefit Ratio of Allogenic Islet Transplantation Under Antithymocyte Globulin-Mycophenolate Mofetil-Tacrolimus Immune Suppression. Transplantation. 2017 Sep;101(9):2218-2227. doi: 10.1097/TP.0000000000001543. PMID 27779572
- [Derived] Ling Z, De Pauw P, Jacobs-Tulleneers-Thevissen D, Mao R, Gillard P, Hampe CS, Martens GA, In't Veld P, Lernmark A, Keymeulen B, Gorus F, Pipeleers D. Plasma GAD65, a Marker for Early beta-Cell Loss After Intraportal Islet Cell Transplantation in Diabetic Patients. J Clin Endocrinol Metab. 2015 Jun;100(6):2314-21. doi: 10.1210/jc.2015-1216. Epub 2015 Mar 27. PMID 25816051
- [Derived] Huurman VA, Hilbrands R, Pinkse GG, Gillard P, Duinkerken G, van de Linde P, van der Meer-Prins PM, Versteeg-van der Voort Maarschalk MF, Verbeeck K, Alizadeh BZ, Mathieu C, Gorus FK, Roelen DL, Claas FH, Keymeulen B, Pipeleers DG, Roep BO. Cellular islet autoimmunity associates with clinical outcome of islet cell transplantation. PLoS One. 2008 Jun 18;3(6):e2435. doi: 10.1371/journal.pone.0002435. PMID 18560516